CLINICAL TRIAL: NCT05773404
Title: Efficacy of Passive Manual Therapy, Active Therapy and Combined Therapy in Relation to the Prevention of Hamstring Injuries in Football Players. Randomised Clinical Trial.
Brief Title: Prevention of Hamstring Injuries in Football Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 313
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Hamstring Injuries
Keywords: physiotherapies techniques; Range of Motion; Hamstring Muscles; Prevention and Control; Muscuoeskeletal Manipulations.
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- passive manual therapy (Experimental): The physiotherapist performs passive techniques on the hamstring muscles of the footballers.
  Interventions: Other: Passive Neurodynamics and Passive axial hip mobilisation/distraction
- active therapy (exercise) (Experimental): The physiotherapist does not perform passive techniques and it is the player who performs active techniques on the hamstring muscles.
  Interventions: Other: Active therapy
- combined therapy (Active Comparator): The physiotherapist performs passive techniques and in addition the player performs active techniques on the hamstring muscles.
  Interventions: Other: 2.5.3. Combined therapy

INTERVENTIONS:
Other: Passive Neurodynamics and Passive axial hip mobilisation/distraction — The physiotherapist performs passive techniques on the hamstring muscles and the nerve that innervates the hamstring muscles.
  Arms: passive manual therapy
Other: Active therapy — Active lumbopelvic CORE control exercises and active stretching of the ischiopelvic nerves
  Other Names: Active Neurodynamics and Therapeutic exercise
  Arms: active therapy (exercise)
Other: 2.5.3. Combined therapy — The physiotherapist performs passive techniques on the hamstring muscles and the nerve that innervates the hamstring muscles and active lumbopelvic CORE control exercises and active stretching of the ischiopelvic nerves.
  Other Names: Passive and Active therapy
  Arms: combined therapy

SUMMARY:
Introduction: The prevalence of hamstring injuries in football is high, causing an increase in the number of casualties and a high socio-economic cost. Currently there are different treatment protocols for this muscle group, but there are often no comparisons of different types of passive, active and combined therapies, and their potential efficacy, in professional football players.

Objectives: To compare the efficacy of three different interventions; passive manual therapy, active therapy based on therapeutic exercise and combined therapy, in relation to hamstring injuries in professional football players.

Methodology: A simple Randomised Clinical Trial (RCT) was conducted (NCT04935398). After applying the selection criteria, a sample of 66 professional football players was obtained. They were divided into 3 intervention groups (A, B and C) with 22 participants in each group and were given passive manual therapy, active therapy (exercise) and combined therapy (sum of the above). The corresponding tests and questionnaires were evaluated to obtain data on hamstring flexibility and hip range of movement at three time periods: pre, post and post2.

ELIGIBILITY:
Inclusion Criteria:

* Professional football athletes.
* Between 18-40 years of age.
* Female gender.
* Active in competitive season.

Exclusion Criteria:

* Neurological signs.
* Inability to follow the evaluator's instructions.
* Physical activity of less than 2 hours per week.
* Serious lower limb injury during the study period.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female footballers
Enrollment: 66 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
range of movements measurements | 1 month
  Observe the degrees of mobility of the lower limb joints.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petersen J, Holmich P. Evidence based prevention of hamstring injuries in sport. Br J Sports Med. 2005 Jun;39(6):319-23. doi: 10.1136/bjsm.2005.018549. PMID 15911599
- [Background] Verrall GM, Slavotinek JP, Barnes PG. The effect of sports specific training on reducing the incidence of hamstring injuries in professional Australian Rules football players. Br J Sports Med. 2005 Jun;39(6):363-8. doi: 10.1136/bjsm.2005.018697. PMID 15911608
- [Result] Hagglund M, Walden M, Ekstrand J. Injury recurrence is lower at the highest professional football level than at national and amateur levels: does sports medicine and sports physiotherapy deliver? Br J Sports Med. 2016 Jun;50(12):751-8. doi: 10.1136/bjsports-2015-095951. Epub 2016 Mar 25. PMID 27015858
- [Result] Ekstrand J, Hagglund M, Walden M. Epidemiology of muscle injuries in professional football (soccer). Am J Sports Med. 2011 Jun;39(6):1226-32. doi: 10.1177/0363546510395879. Epub 2011 Feb 18. PMID 21335353
- [Result] Hagglund M, Walden M, Ekstrand J. Risk factors for lower extremity muscle injury in professional soccer: the UEFA Injury Study. Am J Sports Med. 2013 Feb;41(2):327-35. doi: 10.1177/0363546512470634. Epub 2012 Dec 21. PMID 23263293
- [Result] Ekstrand J, Ueblacker P, Van Zoest W, Verheijen R, Vanhecke B, van Wijk M, Bengtsson H. Risk factors for hamstring muscle injury in male elite football: medical expert experience and conclusions from 15 European Champions League clubs. BMJ Open Sport Exerc Med. 2023 Jan 24;9(1):e001461. doi: 10.1136/bmjsem-2022-001461. eCollection 2023. PMID 36726776
- [Result] Woods C, Hawkins RD, Maltby S, Hulse M, Thomas A, Hodson A; Football Association Medical Research Programme. The Football Association Medical Research Programme: an audit of injuries in professional football--analysis of hamstring injuries. Br J Sports Med. 2004 Feb;38(1):36-41. doi: 10.1136/bjsm.2002.002352. PMID 14751943
- [Result] Arnason A, Andersen TE, Holme I, Engebretsen L, Bahr R. Prevention of hamstring strains in elite soccer: an intervention study. Scand J Med Sci Sports. 2008 Feb;18(1):40-8. doi: 10.1111/j.1600-0838.2006.00634.x. Epub 2007 Mar 12. PMID 17355322